CLINICAL TRIAL: NCT05518149
Title: An Open-label, Long-term, Safety and Efficacy Study of Aticaprant as Adjunctive Therapy in Adult and Elderly Participants With Major Depressive Disorder (MDD)
Brief Title: A Study of Aticaprant in Adult and Elderly Participants With Major Depressive Disorder (MDD)
Acronym: VENTURA-LT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR109218; 67953964MDD3003 (Other: Janssen Research & Development, LLC); 2022-000430-42 (EudraCT Number); 2023-508163-74-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2022-08-25; First posted 2022-08-26 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Depressive Disorder, Major
Keywords: Depressive Disorder, Major; Aticaprant
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Aticaprant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Aticaprant 10 mg (Experimental): Participants will enter this study directly or after completing double-blind phase of studies 67953964MDD3001 or 67953964MDD3002 and will receive Aticaprant 10 milligrams (mg), once daily, orally in addition to the current antidepressant selective serotonin reuptake inhibitor/serotonin-norepinephrine reuptake inhibitor (SSRI/SNRI) therapy on Day 1 up to 52 weeks.
  Interventions: Drug: Aticaprant

INTERVENTIONS:
Drug: Aticaprant — Aticaprant 10 mg tablet will be administered orally.
  Other Names: JNJ-67953964

SUMMARY:
The purpose of this study is to assess the long-term safety and tolerability of aticaprant administered as adjunctive therapy to a current antidepressant (selective serotonin reuptake inhibitor [SSRI] or serotonin and norepinephrine reuptake inhibitor [SNRI]) in all participants with major depressive disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

Transferred-entry participants:

-Participants must have completed the double blind (DB) (expand DB) Treatment Phase of Study 67953964MDD3001 or Study 67953964MDD3002 without early treatment discontinuation or switch in the oral selective serotonin reuptake inhibitor/serotonin-norepinephrine reuptake inhibitor (SSRI/SNRI) in the parent study

Direct-entry participants:

* Have a Hamilton Depression Rating Scale (HDRS)-17 total score of 20 or higher at the first and second screening interviews and must not demonstrate a clinically significant improvement (that is, an improvement of more than 20 percent (%) on their HDRS-17 total score) between the first and the second independent HDRS-17 assessments
* Have had an inadequate response to at least 1 oral antidepressant treatment, administered at an adequate dose (at or above the minimum therapeutic dose per Massachusetts general hospital antidepressant treatment response questionnaire [MGH ATRQ]) and duration (at least 6 weeks) in the current episode of depression
* Must be an outpatient at open-label treatment phase baseline
* Meet Diagnostic and Statistical Manual of Mental Disorders-5th Edition (DSM-5) diagnostic criteria for recurrent or single episode major depressive disorder (MDD), without psychotic features, based upon clinical assessment and confirmed by the Structured Clinical Interview for DSM-5 Axis I Disorders-Clinical Trials Version (SCID-CT)

Direct-entry and Transferred-entry Participants:

-Participants should not take any prohibited medication or food supplements

Exclusion Criteria:

Transferred-entry Participants:

* Participant has been non-compliant with the study intervention administration in the DB Treatment Phase in either of Studies 67953964MDD3001 or 67953964MDD3002 (that is, have missed either 4 or more consecutive doses of study intervention or a total of 8 or more doses during the DB Treatment Phase)
* Participant has any condition or situation/circumstance for which, in the opinion of the investigator, participation would not be in the best interest of the participant (example, compromise the well-being) or that could prevent, limit, or confound the protocol specified assessments

Direct-entry Participants:

* Employee of the investigator or study site, with direct involvement in the proposed study or other studies under the direction of that investigator or study site, as well as family members of the employees or the investigator
* Has a history or evidence of clinically meaningful noncompliance with current antidepressant therapy
* Known allergies, hypersensitivity, or intolerance to aticaprant or any of its excipients

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2025-04-11 (Estimated); Study Completion 2025-04-25 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to Week 54
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have causal relationship with the intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non-investigational) product, whether or not related to that medicinal (investigational or non-investigational) product.
Number of Participants with Adverse Events of Special Interest (AESI) | Up to Week 54
  AEs considered to be of special interest are as Pruritus and Diarrhea.
Number of Participants with Change from Baseline in Vital Signs Abnormalities | Up to Week 54
  Vital signs include body weight, temperature, pulse/heart rate, respiratory rate, pulse oximetry and blood pressure (systolic and diastolic) values.
Number of Participants with Abnormal Body Weight | Up to Week 54
  Participants will be weighed at approximately the same time of day on the same scale, wearing lightweight clothing without shoes; they will be instructed to empty their bladders before being weighed.
Number of Participants with Abnormal Body Mass Index (BMI) | Up to Week 54
  A BMI between 18.5 and 25 kilogram per meter square (kg/m^2) indicates a normal weight.
Percentage of Participants with Suicidal Ideation or Suicidal Behavior based on the Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to Week 54
  C-SSRS is semi structured clinician-administered questionnaire designed to solicit the occurrence, severity, and frequency of suicide-related ideation and behaviors. The maximum score assigned for each participant will also be summarized into one of three categories: no suicidal ideation or behavior (0), suicidal ideation (1-5), suicidal behavior (6-10). Total score ranges from 1 to 10. Higher scores indicate greater severity.
Number of Participants with Abnormalities in Clinical Laboratory parameters | Up to Week 54
  Number of participants with abnormalities in clinical laboratory parameters will be reported.
Number of Participants with Abnormalities in Electrocardiogram (ECG) | Up to Week 54
  Number of participants with abnormalities in ECG will be reported.
Withdrawal Symptoms Assessment Using the Physician Withdrawal Checklist (PWC-20) | Up to Week 54
  Withdrawal symptoms are assessed using the PWC-20. The PWC-20 is a simple and accurate method used to assess potential withdrawal symptoms following cessation of treatment. The PWC-20 is a reliable and sensitive instrument for the assessment of discontinuation symptoms.
Number of participants with Clinically Relevant Sexual Dysfunction Over Time as Measured by the Arizona Sexual Experiences Scale (ASEX) Score | Up to Week 54
  The ASEX is a participant-reported five-item rating scale that quantifies sex drive, arousal, vaginal lubrication/penile erection, ability to reach orgasm, and satisfaction from orgasm. Each of the 5 items is rated on a 6-point scale, ranging from 1 to 6. Total score ranges from 5 to 30, with the higher scores indicating more sexual dysfunction.

SECONDARY OUTCOMES:
Change from Baseline in the Montgomery-asberg Depression Rating Scale (MADRS) Total Score Over Time | Baseline up to Week 54
  Change from baseline in MADRS total score over time will be reported. The MADRS is a clinician-rated scale designed to measure depression severity and detects changes due to antidepressant treatment. The scale consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total score of 60. Higher scores represent a more severe condition.
Change from Baseline in the Participant Health Questionnaire, 9-Item (PHQ-9) Total Score over Time | Baseline up to Week 54
  Change from baseline in PHQ-9 total score over time will be reported. The 9-item PHQ-9 scale scores each of the 9 symptom domains of the Diagnostic and Statistical Manual of Mental Disorders-5th Edition (DSM-5) diagnostic criteria for recurrent or single episode major depressive disorder (MDD) criteria and used both as a screening tool and a measure of response to treatment for depression. Each item is rated on a 4-point scale (0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day). The participant's item responses are summed to provide a total score (range of 0 to 27), with higher scores indicating greater severity of depressive symptoms.
Change from Baseline in Dimensional Anhedonia Rating Scale (DARS) Total Score Over Time | Baseline up to Week 54
  Change from baseline in DARS total score over time will be reported. The DARS is a 17-item self-report questionnaire that is designed to assess anhedonia in MDD, and particularly to increase scale generalizability while maintaining specificity. Respondents provide their own examples of rewarding experiences across the domains of hobbies, social activities, food/drink, and sensory experience. Participants answer a set of standardized questions about desire, motivation, effort and consummatory pleasure with a recall period of "right now" for the examples provided. The instrument is scored as a total sum of all items (range 0-68) with higher scores reflecting increased motivation, effort and pleasure (that is, less anhedonia).
Change from Baseline in the Clinical Global Impression-Severity (CGI-S) Total Score Over Time | Baseline up to Week 54
  Change from baseline in the CGI-S total score over time will be reported. The CGI-S evaluates the severity of psychopathology on a scale of 0 to 7. Considering total clinical experience, a participant is assessed on severity of mental illness at the time of rating according to: 0=not assessed; 1=normal (not at all ill); 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill participants. The CGI-S permits a global evaluation of the participant's condition at a given time.
Percentage of Participants with Greater than or Equal to (>=) 50 percent (%) Reduction from Baseline in the MADRS Total Score Over Time | Week 54
  Percentage of participants with >=50% reduction from baseline in the MADRS total score over time will be reported. The MADRS is a clinician-rated scale designed to measure depression severity and detects changes due to antidepressant treatment. The scale consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total score of 60. Higher scores represent a more severe condition.
Percentage of Participants with Remission of Depressive Symptoms Over Time | Week 54
  Percentage of participants with remission of depressive symptoms over time, defined as a MADRS total score less than or equal to (<=) 10 will be reported. The MADRS is a clinician-rated scale designed to measure depression severity and detects changes due to antidepressant treatment. The scale consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total score of 60. Higher scores represent a more severe condition.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical trial, Study Director — Janssen Research & Development, LLC
Locations (224):
- United States (85):
  - University of Alabama at Birmingham - The Kirklin Clinic, Birmingham, Alabama
  - SW Biomedical Research LLC, Tucson, Arizona
  - University of Arizona, Tucson, Arizona
  - Advanced Research Center Inc, Anaheim, California
  - Proscience Research Group, Culver City, California
  - Behavioral Research Specialists LLC, Glendale, California
  - Sunwise Clinical Research, Lafayette, California
  - Asclepes Research, Long Beach, California
  - Excell Research Inc, Oceanside, California
  - Pacific Neuropsychiatric Specialists, Orange, California
  - Prospective Research Innovations Inc, Rancho Cucamonga, California
  - University of California San Diego Medical Center, San Diego, California
  - Syrentis Clinical Research, Santa Ana, California
  - CMB Clinical Trials, Santee, California
  - California Neuroscience Research, Sherman Oaks, California
  - Viking Clinical Research Ltd, Temecula, California
  - Pacific Clinical Research Medical Group, Upland, California
  - Next Level Clinical Trials, LLC, West Covina, California
  - MCB Clinical Research Centers LLC, Colorado Springs, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - Innovative Research of West Florida, Incorporated, Clearwater, Florida
  - CNS Clinical Research Group, Coral Springs, Florida
  - Gulfcoast Medical Research Center, Fort Myers, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - New Life Medical Research Center, Inc., Hialeah, Florida
  - Amedica Research Institute Inc, Hialeah, Florida
  - Galiz Research, Hialeah, Florida
  - Vertex Clinical Research, Maitland, Florida
  - Vital Care Research, Miami, Florida
  - Global Medical Institutes, Miami, Florida
  - LCC Medical Research Institute Inc, Miami, Florida
  - Pharmax Research Clinic Inc, Miami, Florida
  - A Plus Research, Miami, Florida
  - Florida Research Center Inc., Miami, Florida
  - Ezy Medical Research, Miami, Florida
  - Felicidad Medical Research, Miami, Florida
  - Meridian International Research, Miami Gardens, Florida
  - University of Miami, Miami Lakes, Florida
  - Bravo Health Care Center, North Bay Village, Florida
  - K2 Medical Research, Ocoee, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - APG Research LLC, Orlando, Florida
  - Combined Research Orlando, Orlando, Florida
  - Quantum Laboratories, Pompano Beach, Florida
  - CDC Research Institute LLC, Port Saint Lucie, Florida
  - USF, Department of Psychiatry and Behavioral Neurosciences, Tampa, Florida
  - Research Network America, Berwyn, Illinois
  - Chicago Research Center, Chicago, Illinois
  - Revive Research Institute, Elgin, Illinois
  - Psychiatric Medicine Associates LLC, Skokie, Illinois
  - Tandem Clinical Research, Marrero, Louisiana
  - Clinical Trials of America, Monroe, Louisiana
  - CBH Health, Gaithersburg, Maryland
  - ActivMed Practices and Research, Methuen, Massachusetts
  - Michigan Clinical Research Institute, Ann Arbor, Michigan
  - Psychiatric Care and Research Center (PCRC), O'Fallon, Missouri
  - Midwest Research Group, Saint Charles, Missouri
  - Erie County Medical Center, Buffalo, New York
  - Bioscience Research LLC, Mount Kisco, New York
  - Manhattan Behavioral Medicine, New York, New York
  - Fieve Clinical Research Inc, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Montefiore Medical Center PRIME, The Bronx, New York
  - New Hope Clinical Research, Charlotte, North Carolina
  - Monroe Biomedical Research, Monroe, North Carolina
  - Patient Priority Clinical Sites LLC, Cincinnati, Ohio
  - University of Cincinnati, Dept of Psychiatry & Behavioral Neuroscience, Cincinnati, Ohio
  - Wexner Medical Center at the Ohio State University, Columbus, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Charak Center for Health and Wellness, Garfield Heights, Ohio
  - Conrad Clinical Research, Edmond, Oklahoma
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Paradigm Research Professionals, LLC, Oklahoma City, Oklahoma
  - Lehigh Center for Clinical Research LLC, Allentown, Pennsylvania
  - Suburban Research Associates, Media, Pennsylvania
  - University of Pennsylvania - Perelman School of Medicine, Philadelphia, Pennsylvania
  - Austin Clinical Trial Partners, Austin, Texas
  - West Houston Clinical Research Service, Bellaire, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - North Texas Clinical Trials, Fort Worth, Texas
  - R and H Clinical Research, Katy, Texas
  - Alpine Research Organization, Clinton, Utah
  - Cedar Psychiatry, Murray, Utah
  - University of Virginia, Charlottesville, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
- Argentina (16):
  - INSA Instituto de Neurociencias San Agustín, Buenos Aires
  - STAT Research S A, Buenos Aires
  - CIPREC, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - CENydET - Centro Neurobiologico y de Stress Traumatico, Ciudad Autonoma Buenos Aires
  - CEN Consultorios Especializados en Neurociencias, Córdoba
  - Fundacion Lennox, Córdoba
  - Instituto Medico DAMIC, Córdoba
  - Centro Medico Luquez, Córdoba
  - CENPIA, La Plata
  - Clinica Privada de Salud Mental Santa Teresa de Ávila, La Plata
  - Resolution, Mendoza
  - C I A P Centro de investigacion y Asistencia en Psiquiatria, Rosario
  - Instituto Medico de La Fundacion Estudios Clinicos, Rosario
  - Clinica Mayo de UMCB, San Miguel de Tucumán
  - Clinica El Jardin, Santiago del Estero
- Australia (3):
  - Peninsula Therapeutic & Research Group, Frankston
  - Albert Road Clinic, Melbourne
  - The Alfred Hospital, Melbourne
- Belgium (4):
  - Anima, Alken
  - C.H.U. Brugmann, Brussels
  - Pz Duffel, Duffel
  - Vitaz, Sint-Niklaas
- Brazil (10):
  - Trial Tech Tecnologia em Pesquisas com Medicamentos, Curitiba
  - Universidade Federal do Ceara Hospital Universitario Walter Cantidio, Fortaleza
  - Instituto Goiano de Neuropsiquiatria, Goiânia
  - Associacao Hospitalar Moinhos de Vento, Porto Alegre
  - NPCRS Nucleo de Pesquisa Clinica do Rio Grande do Sul, Porto Alegre
  - Ruschel Medicina e Pesquisa Clínica Ltda, Rio de Janeiro
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos, São Bernardo
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto Hospital de Base, São José do Rio Preto
  - CPQuali Pesquisa Clinica LTDA ME, São Paulo
  - BR Trials, São Paulo
- Bulgaria (11):
  - Ambulatory for Individual Practice for Specialized Medical Care in Psychiatry Dr. Ivo Natsov ET, Cherven Bryag
  - Ambulatory Group practice for specialized help in psychiary Philipopolis ODD, Plovdiv
  - Medical Center Mentalcare OOD, Plovdiv
  - Mental Health Center - Rousse, Rousse
  - Medical Center St. Naum, Sofia
  - MHC - Sofia, EOOD, Sofia
  - DCC 'Sv. Vrach and Sv. Sv. Kuzma and Damyan', OOD, Sofia
  - Medical Center Hera EOOD, Sofia
  - Medical Center Intermedica, OOD, Sofia
  - Diagnostic Consulting Center Mladost - M Varna, Varna
  - Mental Health Center - Veliko Tarnovo EOOD, Veliko Tarnovo
- DIEX Recherche Sherbrooke Inc, Sherbrooke, Quebec, Canada
- China (13):
  - Hebei Mental Health Center, Baoding
  - Beijing Anding Hospital of Capital Medical University, Beijing
  - Peking University Sixth Hospital, Beijing
  - Beijing Huilongguan Hospital, Beijing
  - West China Hospital Sichuan University, Chengdu
  - Guangdong Provincial People's Hospital, Guangzhou
  - Shanghai Mental Health Center, Shanghai
  - Tongji Hospital of Tongji University, Shanghai
  - The First Hospital of Hebei Medical University, Shijiazhuang
  - Tianjin Anding Hospital, Tianjin
  - Wuhan Mental Health Center, Wuhan
  - Wuhu Hospital of Beijing Anding hospital, Wuhu
  - XiAn Mental Healthcare Center, Xi'an
- Czechia (11):
  - Psychiatricka ambulance, MUDr. Marta Holanova, Brno
  - Narodni ustav dusevniho zdravi, Klecany
  - Neuroterapie KH S R O, Kutná Hora
  - A Shine S R O, Pilsen
  - Clintrial s r o, Prague
  - AD71 s.r.o., Prague
  - Praglandia s r o, Prague
  - NeuropsychiatrieHK, s.r.o., Prague
  - Medical Services Prague S R O, Prague
  - Institut Neuropsychiatricke pece, Prague
  - Psychiatricka ordinace, Ústí nad Labem
- France (6):
  - CHU de Brest - Hopital de la Cavale Blanche, Bohars
  - CHU Clermont-Ferrand - Hopital Gabriel Montpied, Clermont-Ferrand
  - Cabinet Medical des Drs Prizac-Desbonnet Scottez, Douai
  - CHU de Nantes hotel Dieu, Nantes
  - Hopital Sainte Anne, Paris
  - CHRU de Tours Clinique Psychiatrique Universitaire, Tours
- Hungary (6):
  - Obudai Egeszsegugyi Centrum Kft, Budapest
  - Semmelweis Egyetem, Budapest
  - Bugat Pal Korhaz, Gyöngyös
  - Dr Mathe es Tarsa Bt, Kalocsa
  - PsychoTech Kft, Pécs
  - Tolna Megyei Balassa Janos Korhaz, Szekszárd
- Italy (7):
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII (Presidio Papa Giovanni XXIII), Bergamo
  - Azienda Ospedaliero Universitaria Mater Domini, Catanzaro
  - AUSL LE di Lecce, Lecce
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - ASST Fatebenefratelli Sacco, Milan
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliera Universitaria Senese Policlinico Santa Maria alle Scotte, Siena
- Poland (8):
  - Mlynowamed Specjalistyczny Psychiatryczny Gabinet Lekarski Joanna Lazarczyk, Bialystok
  - Clinsante Osrodek Badan Klinicznych, Bydgoszcz
  - Centrum Badan Klinicznych PI House sp z o o, Gdansk
  - Centrum Medyczne Care Clinic Katowice, Katowice
  - Specjalistyczna Indywidualna Praktyka Lekarska, Lodz
  - Filip Rybakowski Specjalistyczna Praktyka Lekarska, Poznan
  - Indywidualna Specjalistyczna Praktyka Lekarska Agnieszka Remlinger Molenda, Suchy Las
  - Specjalistyczny Gabinet Psychiatryczny Kowalkowski Gerard, Torun
- Portugal (3):
  - Hospital de Braga, Braga
  - Hospital CUF Inf. Santo, Lisbon
  - Fund. Champalimaud, Lisbon
- Slovakia (8):
  - Psychomed-Svatosavsky, s.r.o., Banská Bystrica
  - Nemocnica s poliklinikou Prievidza so sidlom v Bojniciach, Bojnice
  - Psychiatricka Ambulancia Mentum S.R.O., Bratislava
  - Epamed sro, Košice
  - Univerzitna nemocnica L. Pasteura Kosice, Košice
  - Liptovska Nemocnica S Poliklinikou Mudr. Ivana Stodolu, Liptovský Mikuláš
  - Psychiatricka Ambulancia Psycholine S.R.O., Rimavská Sobota
  - Crystal Comfort s.r.o., Vranov nad Topľou
- South Africa (3):
  - Cape Town Clinical Research Centre, Cape Town
  - Gert Bosch Pretoria South Africa, Pretoria
  - Somerset West Clinical Research Unit, Strand
- South Korea (9):
  - The Catholic University Of Korea St Mary'S Hospital, Bucheon-si
  - Inje University Haeundae Paik Hospital, Busan
  - Korea University Ansan Hospital, Gyeonggi-do
  - Kyung Hee University Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Yeouido St. Mary's Hospital, Seoul
  - Seoul National University Hospital, Seoul
- Spain (10):
  - Institucion Hosp Hestia Palau, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. Univ. La Paz, Madrid
  - Hosp Regional Univ de Malaga, Málaga
  - Hosp. Univ. Son Espases, Palma de Mallorca
  - Hosp. El Bierzo, Ponferrada
  - Corporacio Sanitari Parc Tauli, Sabadell
  - Hosp. Alvaro Cunqueiro, Vigo
  - Hosp. Psiquiatrico Alava, Vitoria-Gasteiz
- Sweden (4):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - ProbarE i Lund AB, Lund
  - ProbarE i Stockholm AB, Stockholm
  - Studieenheten Akademiskt Specialistcentrum Stockholm, Stockholm
- Taiwan (4):
  - China Medical University Hospital, Taichung
  - Taipei Medical University, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Cheng Hsin General Hospital, Taipei
- United Kingdom (2):
  - Institute of Psychiatry, London
  - Moorgreen Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency